CLINICAL TRIAL: NCT02129946
Title: Human Clinical Trial to Investigate the Effects of Resistant Starch Bagels on Risk Factors of Type 2 Diabetes and Colorectal Cancer in Adults at Risk for Type 2 Diabetes
Brief Title: The Effect of Resistant Starch Bagels on Risk Factors of Type 2 Diabetes and Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Collaborators: Ontario Ministry of Agriculture, Food and Rural Affairs (Other Government); Maple Leaf Foods, Canada Bread (Unknown)
Responsible Party: Principal Investigator, Alison Duncan, Alison Duncan, Ph.D., R.D., Professor, University of Guelph
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 13MY041
Record Dates: First submitted 2014-04-29; First posted 2014-05-02 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; Resistant Starch; Postprandial Glucose; Postprandial Insulin; Satiety
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Resistant Starch

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistant Starch Bagels (Active Comparator): Bagels made from high-resistant starch flour (provides 24g resistant starch per day)
  Interventions: Other: Resistant Starch
- Control Bagels (Placebo Comparator): Bagels made from wheat flour
  Interventions: Other: Resistant Starch

INTERVENTIONS:
Other: Resistant Starch — In a randomized crossover fashion, participants will consume bagels that are made with either high-resistant starch or standard wheat flour, daily for a period of 8 weeks, with a 4 week washout period.
  Other Names: RS bagels

SUMMARY:
The purpose of this study is to determine if consumption of bagels made with resistant starch for 8 weeks can improve markers of type 2 diabetes, colon cancer and satiety in adults.

DETAILED DESCRIPTION:
Using a randomized, double-blind crossover study design, we will determine the effect of consuming bagels made with resistant starch daily for 8-weeks can reduce the risk of type 2 diabetes and colon cancer in an adults who are at an increased risk for type 2 diabetes. Additionally, we will compare the satiating effect of these bagels to that of a standard bagel.

ELIGIBILITY:
Inclusion Criteria:

* Males and postmenopausal females at least 40 year old
* BMI ≥25 and <40 kg/m2
* Waist circumference ≥ 102 cm for men, ≥88cm for women
* CANRISK score ≥21 which indicates an elevated risk for type 2 diabetes

Exclusion Criteria:

* Diabetes mellitus (fasting blood glucose ≥ 7.0 mmol/L)
* Restrained eating habits
* Gastrointestinal conditions (Celiac's disease, Crohn's disease, Ulcerative Colitis, Inflammatory Bowel Disease)
* Renal Conditions
* Hepatic Conditions
* Surgery or major medical event within 3 months of study start date
* Select medication use (Glycemia medications, cholesterol-lowering agents, antibiotics within 6 months of the study, other medications known to influence blood glucose insulin, cholesterol, triglycerides, incretin hormones of the digestive tract microbiome)
* Select natural health product (NHP) use (Phytosterols or phytosterol functional foods, other NHPs intended for glycemic or cholesterol control)
* Gluten allergy or intolerance
* Alcohol consumption >15 drinks/week for men and >10 drinks/week for women
* Significant international travel within 6 months of the starting the study, or plans to travel internationally during the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Fasting and postprandial blood glucose | up to day 57 of both treatment periods
  Blood glucose will be measured in the fasting state and postprandially (during a 3-hour oral glucose tolerance test) on the first and last study days of both treatment periods.
Fasting and postprandial insulin | up to day 57 of both treatment periods
  Circulating insulin will be measured in the fasting state and postprandially (during a 3-hour oral glucose tolerance test) on the first and last study days of both treatment periods.

SECONDARY OUTCOMES:
HbA1c | Day 1 and 57 of both treatment periods
  HbA1c (glycated haemoglobin) will be measured from fasting blood drawn on days 1 and 57 of both treatment periods.
Calculated insulin sensitivity and beta-cell function | Days 1 and 57 of both treatment periods
  Data will be used from 3-hour oral glucose tolerance tests performed on days 1 and 57 of both treatment periods.
Satiety-producing effect | Day 2,3 or 4 of both treatment periods
  After study bagel consumption as part of a standard breakfast, questionnaires will be used to quantify subjective measures of satiety, and weighted food records will be used to objectively measure food intake for the rest of the day.

OTHER OUTCOMES:
Sensory response to study bagels | Days 15, 29, 43 and 57 of both treatment periods
  Questionnaires will be used to measure the participants' responses to the aroma, appearance, taste and texture of the study bagels.
Resistant starch bagel tolerance | Days 15, 29, 43 and 57 of both treatment periods
  Questionnaires about bagel tolerance, including subjective ratings of tolerance and any adverse events will be completed every 2 weeks throughout both treatment periods (adverse events will be recorded as often as needed).
Body weight | Days 1, 15, 29, 43 and 57 of both treatment periods
  Body weight will be measures at every study visit.
Fasting serum lipids | On days 1 and 57 of both treatment periods
  Total-cholesterol, LDL-cholesterol, HDL-cholesterol, and triglycerides will be measured from fasted blood samples on days 1 and 57 of both treatment periods.
3-Day food records | Over 3 days during the week before the study start date, and the week before study day 29 of both treatment periods.
  Participants will complete 3-day food records a total of 3 times throughout the study to provide information about their background nutrient intake and dietary habits.

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Duncan, Ph.D., R.D., Study Director — University of Guelph, Human Nutraceutical Research Unit; Alison M Duncan, Ph.D., R.D., Principal Investigator — University of Guelph, Human Nutraceutical Research Unit
Locations (1):
- Human Nutraceutical Research Unit, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Dainty SA, Klingel SL, Pilkey SE, McDonald E, McKeown B, Emes MJ, Duncan AM. Resistant Starch Bagels Reduce Fasting and Postprandial Insulin in Adults at Risk of Type 2 Diabetes. J Nutr. 2016 Nov;146(11):2252-2259. doi: 10.3945/jn.116.239418. Epub 2016 Oct 12. PMID 27733521